CLINICAL TRIAL: NCT00493844
Title: Clinical History and NT-proBNP Versus Exercise Testing for Evaluation of Patients With Acute Chest Pain Without Ischemic Changes in the Electrocardiogram or Troponin Elevation
Brief Title: N-terminal Pro B-type Natriuretic Peptide (Nt-proBNP) Versus Exercise Test for Evaluation of Acute Chest Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Collaborators: Hospital Clinic of Barcelona (Other)
Responsible Party: Principal Investigator, Juan Sanchis, Professor, University of Valencia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 09-27-06
Record Dates: First submitted 2007-06-26; First posted 2007-06-28 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-10

CONDITIONS: Chest Pain
Keywords: Chest pain; Unstable angina; NT-proBNP; Exercise test.
MeSH Terms: conditions — Chest Pain; Angina, Unstable | interventions — Exercise Test; pro-brain natriuretic peptide (1-76)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Discharge if clinical risk score <3 points + Nt-proBNP <110 ng/L
  Interventions: Other: Clinical evaluation + NTproBNP
- 2 (Active Comparator): Discharge if negative exercise testing
  Interventions: Other: Exercise testing

INTERVENTIONS:
Other: Exercise testing — Exercise testing
  Arms: 2
Other: Clinical evaluation + NTproBNP — Clinical evaluation + NTproBNP levels
  Arms: 1

SUMMARY:
The investigators' objective is to compare a new strategy combining clinical history and NT-proBNP levels versus the usual care, consisting of early exercise testing, for decision making in patients presenting to the emergency department with acute chest pain, non-diagnostic electrocardiogram and normal troponin. The investigators hypothesised that the new strategy combining clinical risk score and NT-proBNP will reduce the number of hospitalisations without increasing the number of events during the follow-up.

DETAILED DESCRIPTION:
In patients presenting to the emergency department with acute chest pain, the observation of ischemic changes in the electrocardiogram or troponin elevation prompts hospitalisation and, generally, invasive management. However, decision on admission or discharge is uncertain in the remaining patients. The spectrum of these patients spans from individuals without coronary artery disease to some with high risk unstable angina. An early exercise test is usually performed with the aim of guiding the decision. However, the exercise test is not available 24 hours per day/ 7 days per week, around 40% of the patients show contraindication to exercise and there are inconclusive as well as false-positive results. The limitations of the exercise test can lead to unnecessary hospitalisations. Therefore, there is room for alternative tools. Our objective was to compare a new strategy combining clinical history and NT-proBNP levels versus the usual care, consisting of early exercise testing, for decision making in these patients.

We will randomly compare a new strategy combining a previously published and validated clinical risk score (number of points according to pain characteristics and risk factors) along with NT-proBNP levels, versus the usual strategy using exercise test, for the management of patients presenting to the emergency department with acute chest pain, without ischemia in the electrocardiogram and with normal troponin. In the new strategy, high risk patients (clinical risk score =>3 points) as well as low risk patients (clinical risk score <3 points) but with NT-proBNP >110 ng/L, will be hospitalised; on the other hand, low risk patients (clinical risk score <3 points) with NT-proBNP <110 ng/L will be discharged. In the usual strategy, all patients will be allocated to early exercise test; patients will be hospitalised in case of a positive result, inconclusive result <7 METS or contraindication to exercise, whereas they will be discharged in case of a negative result or inconclusive result with >7 METS without ischemia induction. The primary endpoint will be hospitalisation during the index episode and the secondary endpoints 6-12 months death or acute myocardial infarction, and 6-12month death, myocardial infarction, postdischarge revascularization or readmission by unstable angina.

ELIGIBILITY:
Inclusion Criteria:

* Chest pain of possible coronary origin at criterion of cardiology on duty

Exclusion Criteria:

* Chest pain of obvious non-coronary origin.
* Electrocardiogram showing ST-segment deviation (=>1mm) or T-wave inversion (=>2mm) or atrial fibrillation.
* Troponin elevation at any determination.
* Heart failure at admission.
* Renal failure (creatinine > 1.3 mg/gl).
* Extracardiac disease with life expectancy less than 1 year.
* Structural heart disease different to ischemic heart disease.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 320 (Actual)
Dates: Start 2007-01; Primary Completion 2008-06 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Hospitalization | At the index episode (1 day)

SECONDARY OUTCOMES:
Death, myocardial infarction | 6-12 months
Death, myocardial infarction, postdischarge revascularization or readmission by unstable angina | 6-12 months

CONTACTS AND LOCATIONS:
Overall Officials: Juan Sanchis, MD, Principal Investigator — Hospital Clínico Universitario. Valencia. Spain; Xavier Bosch, MD, Study Chair — Hospital Clínic i Provincial. Barcelona. Spain; Angel Llácer, MD, Study Director — Hospital Clínico Universitario. Valencia. Spain.
Locations (1):
- Hospital Clínico Universitario, Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sanchis J, Bodi V, Nunez J, Bertomeu-Gonzalez V, Gomez C, Bosch MJ, Consuegra L, Bosch X, Chorro FJ, Llacer A. New risk score for patients with acute chest pain, non-ST-segment deviation, and normal troponin concentrations: a comparison with the TIMI risk score. J Am Coll Cardiol. 2005 Aug 2;46(3):443-9. doi: 10.1016/j.jacc.2005.04.037. PMID 16053956
- [Background] Sanchis J, Bodi V, Nunez J, Bertomeu-Gonzalez V, Gomez C, Consuegra L, Bosch MJ, Bosch X, Chorro FJ, Llacer A. Usefulness of early exercise testing and clinical risk score for prognostic evaluation in chest pain units without preexisting evidence of myocardial ischemia. Am J Cardiol. 2006 Mar 1;97(5):633-5. doi: 10.1016/j.amjcard.2005.09.107. Epub 2006 Jan 6. PMID 16490427
- [Background] Sanchis J, Bodi V, Nunez J, Bosch MJ, Bertomeu-Gonzalez V, Consuegra L, Santas E, Gomez C, Bosch X, Chorro FJ, Llacer A. A practical approach with outcome for the prognostic assessment of non-ST-segment elevation chest pain and normal troponin. Am J Cardiol. 2007 Mar 15;99(6):797-801. doi: 10.1016/j.amjcard.2006.10.042. Epub 2007 Jan 30. PMID 17350368
- [Background] Sanchis J, Bosch X, Bodi V, Bellera N, Nunez J, Benito B, Ordonez J, Consuegra L, Heras M, Llecer A. Combination of clinical risk profile, early exercise testing and circulating biomarkers for evaluation of patients with acute chest pain without ST-segment deviation or troponin elevation. Heart. 2008 Mar;94(3):311-5. doi: 10.1136/hrt.2007.115626. Epub 2007 Jul 16. PMID 17639094
- [Result] Sanchis J, Bosch X, Bodi V, Nunez J, Doltra A, Heras M, Mainar L, Santas E, Bragulat E, Garcia-Alvarez A, Carratala A, Llacer A. Randomized comparison between clinical evaluation plus N-terminal pro-B-type natriuretic peptide versus exercise testing for decision making in acute chest pain of uncertain origin. Am Heart J. 2010 Feb;159(2):176-82. doi: 10.1016/j.ahj.2009.11.010. PMID 20152214